CLINICAL TRIAL: NCT06413459
Title: Identification of New Biological Markers for the Progression of Mycobacterium Abscessus-induced Lung Disease in Cystic Fibrosis
Acronym: BioMol-MA
Status: Recruiting | Type: Observational
Sponsor: Ospedale San Raffaele (Other)
Collaborators: Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico (Other)
Responsible Party: Principal Investigator, Nicola Lore, Principal Investigator, Ospedale San Raffaele
Other Study IDs: BioMol-MA
Record Dates: First submitted 2024-05-09; First posted 2024-05-14 (Actual); Last update posted 2024-05-16 (Actual); Status verified 2023-09

CONDITIONS: Non-Tuberculous Mycobacterial Pneumonia; Cystic Fibrosis Lung
Keywords: scRNASec
MeSH Terms: conditions — Cystic Fibrosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — PBMCs and Plasma
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- CF patients with chronic M. abscessus infection
  Interventions: Other: Luminex; scRNAsec
- CF patients with M. abscessus pulmonary disease
  Interventions: Other: Luminex; scRNAsec
- CF patients with no history of M. abscessus infection
  Interventions: Other: Luminex; scRNAsec
- Healty Controls
  Interventions: Other: Luminex; scRNAsec

INTERVENTIONS:
Other: Luminex; scRNAsec — Evaluation of specific cell populations associated with development of M. abscessus lung disease; evaluation of circulating factors related to immunoresponses

SUMMARY:
In this project the investigators aim to identify new biological markers by characterizing the response/inflammation associated with the development and progression of M. abscessus lung disease in patients suffering from cystic fibrosis with the aim of increasing current knowledge available on the development and progression of lung disease.

DETAILED DESCRIPTION:
Main objective:

Evaluate the correlation between early alterations in the profile of specific cell populations or expression markers or soluble immunity activation proteins, considering in particular the development and progression of M. abscessus lung disease in patients with cystic fibrosis.

Secondary objectives

* Identify cellular expression profiles associated with the development and progression of M. abscessus lung disease in cystic fibrosis patients and evaluate its ability to predict clinical outcome
* Identify biomarkers or molecular profiles associated with the development and progression of M. abscessus lung disease in cystic fibrosis patients and evaluate its ability to predict clinical outcome
* Expand pathogenetic knowledge to support disease progression pulmonary disease from M. abscessus in patients with cystic fibrosis and evaluate their ability to predict clinical outcome.
* Describe the reciprocal interactions between cellular and humoral components of the response inflammatory disease during M. abscessus infection with/without M. abscessus lung disease.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a certain diagnosis of cystic fibrosis and visited during normal clinical practice, in accordance with the standard operating procedures in force at the Centres.
* Both sexes
* Age >18 years
* Obtaining informed consent for patients (based on the procedures established by the protocol).

Exclusion Criteria:

* Patients unable to understand the instructions and information provided and be able to adequately accept the study methods.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with cystic fibrosis
Sampling Method: Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2021-04-08 (Actual); Primary Completion 2027-03-30 (Estimated); Study Completion 2027-03-30 (Estimated)

PRIMARY OUTCOMES:
profile of specific cell populations and expression markers to determine the development and progression of M. abscessus lung disease in patients with CF | One month after enrollment visit
  Evaluate the correlation between early alterations in the profile of specific cell populations or expression markers or soluble immunity activation proteins, considering in particular the development and progression of M. abscessus lung disease in patients with cystic fibrosis

CONTACTS AND LOCATIONS:
Locations (1):
- Ospedale San Raffaele, Milan, MI, Italy

IPD SHARING:
Plan to Share IPD: No